CLINICAL TRIAL: NCT06977906
Title: Improved Robotic-Assisted Radical Prostatectomy for Locally Advanced Prostate Cancer: Bladder Suspension and Preliminary Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRCTA,ECFAH of FMU [2025]546
Record Dates: First submitted 2025-05-12; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Robotic-Assisted Radical Prostatectomy; Locally Advanced Prostate Cancer; Bladder Suspension
Keywords: Robotic-Assisted Radical Prostatectomy; Locally Advanced Prostate Cancer; Bladder Suspension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional Robotic Assisted Radical Prostatectomy group (Active Comparator): The conventional RARP utilizes a traditional anterior approach through the patient's head-down, feet-up supine position, with either transabdominal or extraperitoneal access. After establishing pneumoperitoneum, precise dissection of the Retzius space is performed to expose the prostate and surrounding structures. The deep dorsal venous complex is pre-emptively ligated to control bleeding, followed by sharp dissection of the bladder neck while preserving the ureteral orifices. The seminal vesicles and vas deferens are then mobilized, with selective preservation of the neurovascular bundles based on the tumor's characteristics to maintain erectile function. The prostate apex and urethra are delicately dissected while protecting the sphincter, and after complete prostate removal, a continuous, tension-free anastomosis of the bladder and urethra is performed using absorbable sutures. Lymph node dissection is carried out if necessary. Throughout the procedure
  Interventions: Procedure: Improved Robotic-assisted radical prostatectomy group
- Improved Robotic-Assisted Radical Prostatectomy group (Experimental): The procedure is performed in a head-down, feet-up supine position with an abdominal or extraperitoneal approach. The right peritoneum is opened along the right external iliac vein to clear the obturator nerve, vessels, and lymph nodes. The external and internal iliac lymph nodes are also cleared. The right pelvic fascia is incised to remove prostate fat while preserving the bladder's anterior wall peritoneum. The same approach is used on the left side. The peritoneum is retracted to clear anterior prostate fat, and the deep venous complex is ligated to expose the prostate. Prostatectomy is performed, followed by urethra and bladder anastomosis, and peritoneal suturing with drainage tube placement.
  Interventions: Procedure: conventional Robotic-assisted radical prostatectomy group

INTERVENTIONS:
Procedure: conventional Robotic-assisted radical prostatectomy group — Robotic-assisted radical prostatectomy uses a standard anterior approach with transabdominal or extraperitoneal access. After establishing pneumoperitoneum, the Retzius space is dissected to expose the prostate. The deep dorsal venous complex is ligated to control bleeding, and the bladder neck is carefully dissected while preserving the ureters. Seminal vesicles, vas deferens, and neurovascular bundles are selectively preserved based on tumor characteristics. A tension-free anastomosis of the bladder and urethra is performed using absorbable sutures. Lymph node dissection is done if necessary. The robotic system ensures precise dissection, hemostasis, and suturing, optimizing oncological control while preserving urinary continence and sexual function with reduced bleeding and complications.
  Arms: Improved Robotic-Assisted Radical Prostatectomy group
Procedure: Improved Robotic-assisted radical prostatectomy group — The procedure is performed in a head-down, feet-up supine position with an abdominal or extraperitoneal approach. The right peritoneum is opened along the right external iliac vein to clear the obturator nerve, vessels, and lymph nodes. The external and internal iliac lymph nodes are also cleared. The right pelvic fascia is incised to remove prostate fat while preserving the bladder's anterior wall peritoneum. The same approach is used on the left side. The peritoneum is retracted to clear anterior prostate fat, and the deep venous complex is ligated to expose the prostate. Prostatectomy is performed, followed by urethra and bladder anastomosis, and peritoneal suturing with drainage tube placement.
  Arms: conventional Robotic Assisted Radical Prostatectomy group

SUMMARY:
This study is a prospective, single-center clinical trial. It aims to establish an improved robotic-assisted radical prostatectomy for treating locally advanced prostate cancer. The technique evaluates the impact of preserving the anterior peritoneum of the bladder on postoperative bladder descent and urinary control recovery. A retrospective analysis compares this modified approach with traditional anterior approach surgery, assessing differences in oncological outcomes, early functional recovery, and postoperative complication rates. The goal is to provide new theoretical foundations and technical support for the prevention and treatment of postoperative urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. prostate biopsy and clinical confirmation of high-risk prostate cancer (PSA > 20 ng/mL, Gleason score ≥ 8, or cT stage ≥ T2c) followed by robotic-assisted radical prostatectomy
2. multiparametric MRI (mpMRI) with a 3.0 T scanner for prostate or pelvic scans performed within 30 days before the operation at our center
3. Eastern Cooperative Oncology Group (ECOG) performance status score between 0 and 1
4. Complete clinical and prostate biopsy pathological data.
5. General health is good, with no infections, autoimmune diseases, hematologic disorders, or other malignancies.

Exclusion Criteria:

1. Presence of surgical contraindications.
2. refusal of enhanced mpMRI imaging.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
rate of continence | 1 week, 1 month and 3 month after postoperative removal of the urinary catheter
  Time Frame:1 week, 1 month and 3 month after postoperative removal of the urinary catheter
The degree of bladder descent | 1 month after operation
  Time Frame:1 month after operation

CONTACTS AND LOCATIONS:
Locations (1):
- first hospital affiliated of Fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided